CLINICAL TRIAL: NCT05969418
Title: Deep Learning OCT and OCTA Quantification in Neovascular Age Related Macular Degeneration
Brief Title: Deep Learning Optical Coherence Tomography (OCT) and OCT Angiography (OCTA) in NVC
Acronym: OCTA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Doctor, Federico II University
Other Study IDs: 05809850
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Macular Degeneration Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with neovascular macular degeneration
  Interventions: Diagnostic Test: Diagnostic test: using artificial intelligence to evaluate the changes OCT and OCTA parameter
- healty patients matched age and sex without any ocular disease
  Interventions: Diagnostic Test: Diagnostic test: using artificial intelligence to evaluate the changes OCT and OCTA parameter

INTERVENTIONS:
Diagnostic Test: Diagnostic test: using artificial intelligence to evaluate the changes OCT and OCTA parameter — Diagnostic test: using artificial intelligence to evaluate the changes OCT and OCTA parameter before and after ANTI-VEGF treatment

SUMMARY:
To evaluate the activity of neovascular macula degeneretion as assessed by SD-OCTand OCT-A using a split-person study design and deep-learning quantification.

DETAILED DESCRIPTION:
Exudative neovascular macular degeneration is the primarily an age-related retinal condition The optical coherence tomography angiography represents a novel and noninvasive diagnostic technique that allows a detailed and quantitative analysis of retinal and choriocapillary vascular features in order to choose the best therapy .

The study evaluates the changes in structural optical coherence tomography and optical coherence tomography angiography features in neovascular macular degeration patients undergoing ANTI-VEGF treatments using artificial intelligence.

ELIGIBILITY:
Inclusion Criteria: age older than 50 years

* diagnosis of neovascular macular degeneration
* absence of previous retinal surgery and congenital eye diseases.
* absence of errors of refraction
* absence of lens opacities
* absence of low-quality OCT and OCTA images

Exclusion Criteria:• age younger than 50 years

* previous retinal surgery and congenital eye diseases
* errors of refraction
* lens opacities
* low-quality OCT and OCTA images

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 50 years with diagnosis of neovascular macular degeneration. They did not present other ophthalmological disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillary vessel density in patients with macular degeneration complicated by nvc | more than sixmonths

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, MD, Study Chair — Federico II University
Locations (1):
- Federico II University, Naples, Italy